CLINICAL TRIAL: NCT01968213
Title: A Study of Rucaparib as Switch Maintenance Following Platinum-Based Chemotherapy in Patients With Platinum-Sensitive, High-Grade Serous or Endometrioid Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Cancer ( ARIEL3 )
Brief Title: Phase 3 Study of Rucaparib as Switch Maintenance After Platinum in Relapsed High Grade Serous or Endometrioid Ovarian Cancer (ARIEL3)
Acronym: ARIEL3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Collaborators: Foundation Medicine (Industry); Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CO-338-014; 2013-000518-39 (EudraCT Number)
Record Dates: First submitted 2013-10-17; First posted 2013-10-23 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: ARIEL3; ARIEL 3; platinum sensitive; PARP Inhibitor; rucaparib; homologous recombination; homologous recombination deficiency; CO-338; PF 01367338; AG 14699; platinum sensitive ovarian cancer; platinum sensitive fallopian tube cancer; platinum sensitive primary peritoneal cancer; platinum sensitive peritoneal cancer; gynecological cancer; Clovis; Clovis Oncology
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — rucaparib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rucaparib (Experimental): Oral tablets administered twice daily with 8 oz (240 mL) of water on an empty stomach or with food; 28-day cycles of treatment. Doses should be taken as close to 12 hours apart as possible, preferably at the same times every day. Tablets should be swallowed whole.
  Interventions: Drug: Rucaparib
- Placebo (Placebo Comparator): Oral tablets administered twice daily with 8 oz (240 mL) of water on an empty stomach or with food; 28-day cycles of treatment. Doses should be taken as close to 12 hours apart as possible, preferably at the same times every day. Tablets should be swallowed whole.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rucaparib — Oral tablets administered twice daily with 8 oz (240 mL) of water on an empty stomach or with food; 28-day cycles of treatment. Doses should be taken as close to 12 hours apart as possible, preferably at the same times every day. Tablets should be swallowed whole.
  Other Names: CO-338; PF 01367338; AG 14699
  Arms: Rucaparib
Drug: Placebo — Oral tablets administered twice daily with 8 oz (240 mL) of water on an empty stomach or with food; 28-day cycles of treatment. Doses should be taken as close to 12 hours apart as possible, preferably at the same times every day. Tablets should be swallowed whole.
  Arms: Placebo

SUMMARY:
Patients enrolled into this study will be stratified into 3 groups based on gene mutations identified in their tumor tissue. The purpose of this study is to evaluate patient response to maintenance treatment with rucaparib versus placebo. Response to treatment will be analyzed based on homologous recombination (HR) status of tumor samples.

DETAILED DESCRIPTION:
Rucaparib is an orally available, small molecule inhibitor of poly-adenosine diphosphate [ADP] ribose polymerase (PARP) being developed for treatment of ovarian cancer associated with homologous recombination (HR) DNA repair deficiency (HRD). Clinical data have shown that ovarian cancer patients with and without evidence of a gBRCA mutation benefit from treatment with a PARP and that maintenance treatment with a PARP inhibitor following a response to platinum-based treatment increases PFS in patients with ovarian cancer. While patients with a BRCA mutation derived the most benefit, patients without evidence of a BRCA mutation also derived significant benefit.

Patients enrolled into this study will be stratified into 3 groups based on tumor HRD status. The purpose of this study is to identify which of these groups of patients will most likely benefit from treatment with rucaparib. It is anticipated that rucaparib will provide therapeutic benefit and increase PFS in patients with HRD associated with a BRCA gene mutation or other HR gene alteration.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of high-grade serous or endometrioid epithelial ovarian, primary peritoneal, or fallopian tube cancer.
* Received ≥2 prior platinum-based treatment regimens including platinum based regimen that must have been administered immediately prior to maintenance therapy in this trial.
* Received no more than 1 non-platinum chemotherapy regimen. Prior hormonal therapy will not be counted as a non-platinum regimen.
* Must have had at least a 6-month disease-free period following prior treatment with the penultimate platinum-based chemotherapy and achieved a response.
* For the last chemotherapy course prior to study entry, patients must have received a platinum-based doublet chemotherapy regimen and have achieved a CR or PR (as defined by RECIST) and/or a GCIG CA-125 response.
* Have sufficient archival tumor tissue for analysis.

Exclusion Criteria:

* History of prior cancer except for non-melanoma skin cancer, breast cancer curatively > 3 years ago, curatively treated solid tumor (>5 years ago without evidence of recurrence), and synchronous endometrial cancer (Stage 1A) with ovarian cancer.
* Prior treatment with any PARP inhibitor, including rucaparib. Patients who received prior iniparib are eligible.
* Untreated or symptomatic central nervous system metastases.
* Pre-existing duodenal stent and/or any gastrointestinal disorder or defect that would, in the opinion of the Investigator, interfere with absorption of study drug.
* Required drainage of ascites during the final 2 cycles of their last platinum-based regimen and/or during the period between the last dose of chemotherapy of that regimen and randomization to maintenance treatment in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Giordano, Study Director — Clovis Oncology, Inc.
Locations (96):
- United States (22):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Saint Jude Heritage Medical Center, Fullerton, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Central Coast Medical Oncology, Santa Maria, California
  - University of California Los Angeles (UCLA), Santa Monica, California
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Memorial Healthcare System, Hollywood, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Johns Hopkins Universty, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute - Wayne State University, Detroit, Michigan
  - Washington University School of Medicine - Division of Gynaecological Oncology, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hope Women's Cancer Centers, Asheville, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington at Seattle, Seattle, Washington
- Australia (7):
  - Prince of Wales Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - St John of God Hospital Subiaco, Subiaco, Western Australia
- Belgium (4):
  - AZ St Augustinus, Antwerp
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Clinique Sainte-Elisabeth, Namur
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec, Québec
- France (9):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Centre Francois Baclesse, Caen, Basse-Normandie
  - Institut Claudius Regaud, Toulouse, Midi-Pyrenees
  - Centre Catherine de Sienne, Nantes, Pays de la Loire Region
  - Institute Bergonie, Bordeaux
  - Hospital Tenon, Paris
  - Hôpital Européen Georges-Pompidou, Paris, Île-de-France Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Germany (7):
  - Klinikum Ludwigsburg-Bietigheim gGmbH, Ludwigsburg, Baden-Wuerttembert
  - Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Rotkreuzklinikum Muenchen gGmbH, Munich, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Dr. Horst Schmidt Klinik, Klinik fuer Gynaekologie und Gyn. Onkologie, Wiesbaden, Hesse
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Technische Universität Dresden, Dresden, Saxony
- Israel (6):
  - Rambam Health Care Campus, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Oncology Institute, Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh M.C., Ẕerifin
- Italy (8):
  - Oncology Unit City Hospital degli Infermi, Faenza, Ravenna
  - Arcispedale Santa Maria Nuova IRCCS, Reggio Emilia, Reggio Nella Emilia
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Fondazione IRCCS National Cancer Institute, Milan
  - Instituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero Universitaria Policlinico di Modena, Modena
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Policlinico Universitario Agostino Gemelli, Roma
- New Zealand (3):
  - Auckland City Hospital, Auckland, Grafton
  - Palmsteron North Hospital, Palmerston North, Manawatu
  - Wellington Hospital, Newtown, Wellington Region
- Spain (10):
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Centro Oncologico de Galica, A Coruña
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Centro Integral Oncológico Clara Campal, Hospital de Madrid Norte-San Chinarro, Madrid
  - Hospital Regional Universitario Carlos Haya de Malaga, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Valencia de Oncologia-Fundacion, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (12):
  - Royal Marsden Hospital, London, England
  - Belfast City Hospital, Belfast, Northern Ireland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - St. James University Hospital, Leeds, West Yorkshire
  - Addenbrookes Hospital, Cambridge
  - Barts Health NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Sarah Cannon Reserach Institute UK, London
  - University College London, London
  - The Christie NHS Foundation Trust, Manchester
  - Sir Bobby Robson Cancer trials research Centre, Northern Centre For Cancer Care, Newcastle upon Tyne

REFERENCES:
- [Derived] Peipert JD, Goble S, Isaacson J, Tang X, Wallace K, Coleman RL, Ledermann JA, Cella D. Patient-reported outcomes of maintenance rucaparib in patients with recurrent ovarian carcinoma in ARIEL3, a phase III, randomized, placebo-controlled trial. Gynecol Oncol. 2023 Aug;175:1-7. doi: 10.1016/j.ygyno.2023.05.060. Epub 2023 May 30. PMID 37262961
- [Derived] Green ML, Ma SC, Goble S, Giordano H, Maloney L, Simmons AD, Beltman J, Harding TC, Xiao JJ. Population pharmacokinetics of rucaparib in patients with advanced ovarian cancer or other solid tumors. Cancer Chemother Pharmacol. 2022 May;89(5):671-682. doi: 10.1007/s00280-022-04413-7. Epub 2022 Apr 10. PMID 35397664
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- [Derived] Colombo N, Oza AM, Lorusso D, Aghajanian C, Oaknin A, Dean A, Weberpals JI, Clamp AR, Scambia G, Leary A, Holloway RW, Gancedo MA, Fong PC, Goh JC, O'Malley DM, Armstrong DK, Banerjee S, Garcia-Donas J, Swisher EM, Meunier J, Cameron T, Maloney L, Goble S, Bedel J, Ledermann JA, Coleman RL. The effect of age on efficacy, safety and patient-centered outcomes with rucaparib: A post hoc exploratory analysis of ARIEL3, a phase 3, randomized, maintenance study in patients with recurrent ovarian carcinoma. Gynecol Oncol. 2020 Oct;159(1):101-111. doi: 10.1016/j.ygyno.2020.05.045. Epub 2020 Aug 26. PMID 32861537
- [Derived] Ledermann JA, Oza AM, Lorusso D, Aghajanian C, Oaknin A, Dean A, Colombo N, Weberpals JI, Clamp AR, Scambia G, Leary A, Holloway RW, Gancedo MA, Fong PC, Goh JC, O'Malley DM, Armstrong DK, Banerjee S, Garcia-Donas J, Swisher EM, Cameron T, Maloney L, Goble S, Coleman RL. Rucaparib for patients with platinum-sensitive, recurrent ovarian carcinoma (ARIEL3): post-progression outcomes and updated safety results from a randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2020 May;21(5):710-722. doi: 10.1016/S1470-2045(20)30061-9. PMID 32359490
- [Derived] Coleman RL, Oza AM, Lorusso D, Aghajanian C, Oaknin A, Dean A, Colombo N, Weberpals JI, Clamp A, Scambia G, Leary A, Holloway RW, Gancedo MA, Fong PC, Goh JC, O'Malley DM, Armstrong DK, Garcia-Donas J, Swisher EM, Floquet A, Konecny GE, McNeish IA, Scott CL, Cameron T, Maloney L, Isaacson J, Goble S, Grace C, Harding TC, Raponi M, Sun J, Lin KK, Giordano H, Ledermann JA; ARIEL3 investigators. Rucaparib maintenance treatment for recurrent ovarian carcinoma after response to platinum therapy (ARIEL3): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Oct 28;390(10106):1949-1961. doi: 10.1016/S0140-6736(17)32440-6. Epub 2017 Sep 12. PMID 28916367
- See also: ARIEL program website — http://www.arielstudy.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 564 subjects were recruited from 87 sites across 11 countries and randomized (2:1) to treatment with rucaparib or placebo
Groups:
- Rucaparib 600 mg Tablets; Placebo Tablets: Taken orally twice daily (continuous 28 day treatment cycles)
Period: Overall Study
Arm/Group | Rucaparib 600 mg Tablets | Placebo Tablets
Started | 375 | 189
Completed | 375 | 189
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rucaparib 600 mg Tablets | Placebo Tablets | Total
Number analyzed (Participants) | 375 | 189 | 564
Age, Continuous [Median (Full Range); unit: Years] | 61 [39 to 84] | 62 [36 to 85] | 61 [36 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 375 | 189 | 564
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 14 | 7 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 292 | 144 | 436
  More than one race | 12 | 8 | 20
  Unknown or Not Reported | 48 | 27 | 75
Best Response from Previous Platinum Therapy [Count of Participants; unit: Participants] — Complete and partial responses at baseline must have been reported according to RECIST v1.1, as assessed by CT/MRI, and GCIG CA-125 response criteria, and defined as: Complete Response (CR) i.e. absence of any detectable disease and CA-125<ULN; Partial Response (PR), ≥30% decrease in the sum of the longest diameter of measurable lesions or if non-measurable disease at baseline, a GCIG CA-125 response (least a 50% reduction in CA-125 levels from a pretreatment sample (which must have initially been 2xULN) and confirmed after ≥21 days). CA-125 must have been <ULN for all PRs.
  Participants
    RECIST CR | 126 | 64 | 190
    RECIST / CA-125 PR | 249 | 125 | 374
Penultimate Progression-free (PF) Interval [Count of Participants; unit: Participants] — Progressive disease is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of measurable lesions, an unequivocal increase in existing non-measurable lesion(s), or the appearance of unequivocal new lesion(s).
  Participants
    6-12 Months | 151 | 76 | 227
    >12 Months | 224 | 113 | 337
Bulky Lesions (lesion >20 mm) at Baseline [Count of Participants; unit: Participants]
  Yes | 71 | 29 | 100
  No | 304 | 160 | 464

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression According to RECIST Version 1.1, as Assessed by the Investigator, or Death From Any Cause (Investigator Progression Free Survival as Per invPFS)
Description: Progression-free survival by Investigator (invPFS) is defined as the time from randomization to disease progression, according to RECIST v1.1 criteria as assessed by the investigator, or death due to any cause, whichever occurs first. Progressive disease is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of measurable lesions, an unequivocal increase in existing non-measurable lesion(s), or the appearance of unequivocal new lesion(s).
Time Frame: Every 12 calendar weeks (within 7 days prior is permitted) after start of treatment until treatment discontinuation due to disease progression. Total follow-up was up to approximately 3 years.
Population: Intent-to-treat: All patients randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rucaparib 600 mg Tablets | Placebo Tablets
Number analyzed (Participants) | 375 | 189
Months | 10.8 [8.3 to 11.4] | 5.4 [5.3 to 5.5]
Statistical Analysis 1: Comparison: Rucaparib 600 mg Tablets vs Placebo Tablets; Test type: Superiority; p < 0.0001, Regression, Cox; Cox Proportional Hazard = 0.365, 95% CI 2-sided [0.295 to 0.451]; Analysis is performed by randomization strata of HRD classification by CTA, best response, and penultimate platinum progression-free interval

2. Secondary Outcome: Disease Progression According to RECIST v1.1, as Assessed by Independent Radiology Review (IRR), or Death From Any Cause (irrPFS)
Description: To evaluate PFS by RECIST v1.1, as assessed by independent radiology review (IRR).
Time Frame: Every 12 calendar weeks (within 7 days prior is permitted) after start of treatment until treatment discontinuation due to disease progression. Total follow-up was up to approximately 8.2 years.
Population: Intent-to-treat: All patients randomized
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib 600 mg Tablets | Placebo Tablets
Number analyzed (Participants) | 375 | 189
months | 13.7 [11.0 to 19.1] | 5.4 [5.1 to 5.5]
Statistical Analysis 1: Comparison: Rucaparib 600 mg Tablets vs Placebo Tablets; Test type: Superiority; p < 0.0001, Regression, Cox; Cox Proportional Hazard = 0.354, 95% CI 2-sided [0.278 to 0.450]; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the number of days from the date of randomization to the date of death (due to any cause). Patients who are still alive were censored on the date of their last available visit or last date known to be alive.
Time Frame: All patients were followed for survival up to approximately 8.2 years.
Population: Intent-to-treat: All patients randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rucaparib 600 mg Tablets | Placebo Tablets
Number analyzed (Participants) | 375 | 189
Months | 36.0 [32.8 to 39.4] | 43.2 [38.1 to 46.9]

4. Secondary Outcome: Time to a 4-point Decrease in the Disease-related Symptoms - Physical (DRS-P) Subscale of the FOSI-18
Description: The National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy (NCCN-FACT) FACT-Ovarian Symptom Index (FOSI-18) is a questionnaire, for completion by patients, designed to assess the impact of cancer therapy on ovarian cancer-related symptoms and is based on numerical point scoring of symptoms. The DRS-P subscale of the questionnaire is specifically designed to assess physical symptoms of ovarian cancer and evaluate changes in the subscale point score in individual assessments over time. This study looked at the time to a 4-point reduction in subscale score as an indicator of improvement in disease-related physical symptoms on cancer therapy.
Time Frame: Screening, Day 1 of each treatment cycle, Treatment Discontinuation visit, and 28-day Follow-up visit. Total follow-up was up to approximately 6.4 years.
Population: Intent-to-treat: All patients randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rucaparib 600 mg Tablets | Placebo Tablets
Number analyzed (Participants) | 375 | 189
Months | 1.9 [1.8 to 2.8] | 6.4 [4.6 to 9.2]

5. Secondary Outcome: Time to an 8-point Decrease in the Total Score of the FOSI-18
Description: The National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy (NCCN-FACT) FACT-Ovarian Symptom Index (FOSI-18) is a questionnaire, for completion by patients, designed to assess the impact of cancer therapy on ovarian cancer-related physical, emotional and treatment-related symptoms, and is based on numerical point scoring of symptoms. The questionnaire is designed to evaluate changes in the total score in individual assessments over time. This study looked at the time to an 8-point reduction in the total score as an indicator of improvement in disease-related symptoms on cancer therapy.
Time Frame: as for outcome 4
Population: Intent-to-treat: All patients randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rucaparib 600 mg Tablets | Placebo Tablets
Number analyzed (Participants) | 375 | 189
Months | 2.9 [2.7 to 3.7] | 10.8 [9.2 to 17.5]

6. Secondary Outcome: Individual Model Parameter Estimates of Rucaparib and Covariates Identification
Description: Concentration summary statistics
Time Frame: Study data collection occurred over approximately 7 months.
Population: All patients who are treated with rucaparib with at least one pharmacokinetic (PK) measurement
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Rucaparib 600 mg Tablets
Number analyzed (Participants) | 295
ng/mL
  Cycle 2 Day 1 | 1128 (95.42)
  Cycle 4 Day 1 | 1136 (86.19)
  Cycle 7 Day 1 | 1165 (78.53)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date of first dose of study drug and until 28 days after last dose of study drug, approximately 8.2 years.
Description: Three patients were randomized to the rucaparib arm and discontinued prior to receiving study drug.
  Reasons for discontinuation were due to withdrawal of consent, physician decision, and laboratory value (did not meet eligibility criteria)
Arm/Group | Rucaparib 600 mg Tablets | Placebo Tablets
All-Cause Mortality (participants affected / at risk) | 9/372 | 2/189
Serious Adverse Events (participants affected / at risk) | 91/372 | 20/189
Other Adverse Events (participants affected / at risk) | 372/372 | 182/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib 600 mg Tablets (N=372) | Placebo Tablets (N=189)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 3 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 9 | 2
General physical health deterioration (General disorders) | 2 | 0
Incarcerated hernia (General disorders) | 2 | 0
Pyrexia (General disorders) | 6 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0
Stoma site infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Varicella (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 0
Gastrointestinal stoma output increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell unclassifiable lymphoma high grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 18 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 3 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Behaviour disorder (Psychiatric disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib 600 mg Tablets (N=372) | Placebo Tablets (N=189)
Abdominal distension (Gastrointestinal disorders) | 49 | 22
Abdominal pain (Gastrointestinal disorders) | 121 | 50
Abdominal pain upper (Gastrointestinal disorders) | 57 | 11
Constipation (Gastrointestinal disorders) | 143 | 44
Diarrhoea (Gastrointestinal disorders) | 130 | 43
Dry mouth (Gastrointestinal disorders) | 30 | 9
Dyspepsia (Gastrointestinal disorders) | 58 | 9
Nausea (Gastrointestinal disorders) | 284 | 70
Stomatitis (Gastrointestinal disorders) | 35 | 5
Vomiting (Gastrointestinal disorders) | 140 | 29
Mucosal inflammation (General disorders) | 34 | 9
Oedema peripheral (General disorders) | 43 | 16
Pyrexia (General disorders) | 54 | 9
Influenza (Infections and infestations) | 32 | 4
Nasopharyngitis (Infections and infestations) | 38 | 12
Sinusitis (Infections and infestations) | 20 | 3
Upper respiratory tract infection (Infections and infestations) | 48 | 6
Urinary tract infection (Infections and infestations) | 39 | 9
Blood alkaline phosphatase increased (Investigations) | 22 | 1
Blood creatinine increased (Investigations) | 64 | 3
Weight decreased (Investigations) | 30 | 3
White blood cell count decreased (Investigations) | 26 | 8
Decreased appetite (Metabolism and nutrition disorders) | 94 | 25
Hypercholesterolaemia (Metabolism and nutrition disorders) | 28 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 44 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 81 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 57 | 26
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 17
Dizziness (Nervous system disorders) | 61 | 15
Dysgeusia (Nervous system disorders) | 114 | 11
Headache (Nervous system disorders) | 74 | 31
Anxiety (Psychiatric disorders) | 31 | 14
Depression (Psychiatric disorders) | 33 | 6
Insomnia (Psychiatric disorders) | 58 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 67 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 57 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 36 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 39 | 16
Erythema (Skin and subcutaneous tissue disorders) | 32 | 5
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 69 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 54 | 22
Rash (Skin and subcutaneous tissue disorders) | 54 | 17
Hot flush (Vascular disorders) | 23 | 8
Hypertension (Vascular disorders) | 43 | 16
Anaemia (Blood and lymphatic system disorders) | 139 | 9
Neutropenia (Blood and lymphatic system disorders) | 51 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 65 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 21 | 7
Asthenia (General disorders) | 87 | 20
Fatigue (General disorders) | 192 | 66
Influenza like illness (General disorders) | 22 | 2
Alanine aminotransferase increased (Investigations) | 129 | 4
Aspartate aminotransferase increased (Investigations) | 102 | 3
Neutrophil count decreased (Investigations) | 31 | 6
Platelet count decreased (Investigations) | 52 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 21 | 5
Taste disorder (Nervous system disorders) | 38 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 26 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT01968213/Prot_002.pdf
  • Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT01968213/SAP_001.pdf